CLINICAL TRIAL: NCT02605954
Title: A Phase 3b, Randomized, Open-Label Study to Evaluate the Safety and Efficacy of Switching From Regimens Consisting of Abacavir/Lamivudine (ABC/3TC) Plus a Third Antiretroviral Agent to the Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) Fixed-Dose Combination (FDC) in Virologically-Suppressed HIV 1 Infected Adult Subjects
Brief Title: Safety and Efficacy of Switching From Regimens of ABC/3TC + a 3rd Agent to E/C/F/TAF Fixed-Dose Combination (FDC) in Virologically-Suppressed HIV 1 Infected Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-292-1823; 2015-002711-15 (EudraCT Number)
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-06

CONDITIONS: HIV-1 Infection
Keywords: HIV 1 Infection; HIV; Virologically-Suppressed; Antiretroviral agents
MeSH Terms: interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; abacavir, lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- E/C/F/TAF (Experimental): Participants will switch to E/C/F/TAF FDC and receive treatment for 48 weeks.
  Interventions: Drug: E/C/F/TAF
- ABC/3TC+3rd Agent (Active Comparator): Participants will maintain prior regimen of ABC/3TC plus a third antiretroviral agent for 24 weeks followed by a delayed switch to E/C/F/TAF FDC.
  Note: the prior regimen is determined by the participant's clinician (prior to entry into the study) and will consist of one of the third antiretroviral agents listed.
  Interventions: Drug: ABC/3TC; Drug: Third Antiretroviral Agent

INTERVENTIONS:
Drug: E/C/F/TAF — 150/150/200/10 mg FDC tablets administered orally once daily
  Other Names: Genvoya®
  Arms: E/C/F/TAF
Drug: ABC/3TC — 600/300 mg tablets administered orally once daily
  Other Names: Epzicom; Kivexa
  Arms: ABC/3TC+3rd Agent
Drug: Third Antiretroviral Agent — Third antiretroviral agents could include one of the following:
  * ATV+cobicistat (COBI; Tybost®) or ATV/COBI FDC
  * DRV+COBI or DRV/COBI FDC
  * darunavir (DRV; Prezista®) + RTV
  * lopinavir/ritonavir (LPV/r; Kaletra®)
  * atazanavir (ATV; Reyataz®) + ritonavir (RTV; Norvir®)
  * efavirenz (EFV; Sustiva®)
  * etravirine (ETR; Intelence®)
  * nevirapine (NVP; Viramune®)
  * rilpivirine (RPV; Edurant®)
  * dolutegravir (DTG; Tivicay®)
  * raltegravir (RAL; Isentress®)
  * fosamprenavir (FPV; Lexiva®) + RTV
  * saquinavir (SQV; Invirase®) + RTV
  * ATV (no booster)
  Drug classes:
  * Protease inhibitors (PI): LPV/r, ATV, RTV, ATV, DRV, FPV and SQV
  * Pharmacokinetic enhancer: COBI
  * Non-nucleoside reverse transcriptase inhibitors (NNRTI): EFV, RPV, NVP, and ETR
  * Integrase inhibitors: RAL and DTG
  Arms: ABC/3TC+3rd Agent

SUMMARY:
The primary objective of this study is to evaluate the efficacy of switching to elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) fixed-dose combination (FDC) relative to continuing on a baseline regimen consisting of abacavir/lamivudine (ABC/3TC) plus a 3rd antiretroviral agent in HIV-1 infected participants.

ELIGIBILITY:
Key Inclusion Criteria:

HIV-infected adult participants who meet the following criteria will be given the option to participate in the study:

* Currently receiving ABC/3TC plus a third antiretroviral (ARV) agent for ≥ 6 consecutive months preceding the screening visit. For subjects with 3 or more ART regimens, a regimen history must be provided to the Sponsor for approval. Allowed third antiretroviral agents include LPV/r, ATV+RTV, ATV+COBI (or ATV/COBI FDC), DRV+RTV, DRV + COBI (or DRV/COBI FDC) FPV + RTV, SQV + RTV, ATV (no booster), EFV, RPV, NVP, ETR, RAL or DTG
* Documented plasma HIV-1 RNA levels < 50 copies/mL for ≥ 6 months preceding the screening visit (measured at least twice using the same assay). In the preceding 6 months prior to screening, one episode of "blip" (HIV-1 RNA > 50 and < 400 copies/mL) is acceptable, only if HIV-1 RNA is < 50 copies/mL immediately before and after the "blip".
* Plasma HIV-1 RNA < 50 copies/mL at screening visit
* Individuals will have no evidence of previous virologic failure on a PI+RTV or integrase strand transfer inhibitor-based regimen (with or without resistance to either class of ARV).
* All documented historical plasma genotype(s) must not show resistance to tenofovir disoproxil fumarate (TDF) or emtricitabine (FTC), including, but not limited to the presence of reverse transcriptase resistance mutants K65R, K70E, M184V/I, or thymidine analog associated mutations (TAMs) (TAMs are: M41L, D67N, K70R, L210W, T215Y/F, K219Q/E/N/R). If a historical genotype is not available or subject has 3 or more ART regimens, subject will have proviral genotype analysis prior to Day 1 to confirm absence of archived resistance to TDF or FTC.
* Adequate renal function defined as having an estimated glomerular filtration rate of ≥ 30 mL/min as calculated by Cockcroft-Gault (eGFR-CG)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2018-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (49):
- United States (12):
  - Spectrum Medical Group, Phoenix, Arizona
  - Ruane Clinical Research Group, Los Angeles, California
  - Capital Medical Associates, P.C., Washington D.C., District of Columbia
  - Georgetown University, Washington D.C., District of Columbia
  - Gary Richmond, MD, PA, Inc., Fort Lauderdale, Florida
  - Midway Immunology & Research Center, LLC, Ft. Pierce, Florida
  - Steinhart Medical Associates dba The Kinder Medical Group, Miami, Florida
  - Triple O Research Institute PA, West Palm Beach, Florida
  - The Positive Health Clinic, Allegheny Health Network, Pittsburgh, Pennsylvania
  - Central Texas Clinical Research, Austin, Texas
  - AIDS Arms, Inc./Trinity Health & Wellness Center, Dallas, Texas
  - Tarrant County ID Associates, Fort Worth, Texas
- France (11):
  - CHU - Groupe Saint-Andre, Bordeaux
  - Hopital Henri Mondor, Créteil
  - Hopital Europeen Marseille, Marseille
  - C.H.U. de Nantes, Nantes
  - C.H.U. de NICE, Nice
  - CHU Hotel Dieu, Paris
  - Hopital Lariboisiere, Paris
  - Hopital Necker les Enfants Malades, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Gustave Dron, Tourcoing
- Germany (4):
  - Epimed GmbH, Berlin
  - Universitatsklinikum Essen, Essen
  - ICH Study Center Hamburg, Hamburg
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
- Italy (11):
  - ARNAS Garibaldi - Nesima, Catania
  - Unit Infectious Diseases - University of Catania - ARNAS Garibaldi, Catania
  - Azienda Ospedaliera Luigi Sacco, Milan
  - Azienda Ospedaliero Universitaria Policlinico di Modena, Modena
  - Azienda Ospedale San Paolo, Monza
  - Azienda Ospedaliera San Gerardo, Monza
  - Ospedale Civile S. Spirito AUSL, Pescara
  - Unità Operativa Complessa di Malattie Infettive, Pescara
  - Istituto Nazionale Malattie Infettive Lazzaro Spallanzani I.R.C.C.S., Roma
  - Comprensorio Ospedaliero Amedeo di Savoia, Torino
  - Dipartimento di Malattie Infettive e Tropicali, Torino
- Spain (10):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Costa Del Sol, Marbella
  - Hospital Reg. Univ. Carlos Haya, Málaga
  - Hospital Clínico Universitario de Valencia (Galindo), Valencia
  - Hospital General Universitario de Valencia (Abril), Valencia
  - Hospital Alvaro Cunqueiro, Vigo
- Mortimer Market Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Background] A Gori, G Rizzardini, C Miralles, J Olalla, JM Molina, F Raffi, P Kumar, A Antinori, M Ramgopal, HJ Stellbrink, M Das, H Chu, R Ram, W Garner, SK Chuck, D Piontkowsky, R Haubrich. Switching from An Abacavir (ABC)/Lamivudine (3TC)-Based Regimen to a Single-Tablet Regimen of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) is Efficacious and Safe: Week 24 Primary Analysis of a Randomized Controlled Study in Virologically-Suppressed Adults [Presentation]. XVIII Congrès National de la SFLS, 19-20 October 2017, Nice Acropolis, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe and North America. The first participant was screened on 18 November 2015. The last study visit occurred on 24 Jan 2018.
Pre-assignment Details: 346 participants were screened.
Groups:
- E/C/F/TAF: Elvitegravir/ cobicistat/ emtricitabine/tenofovir alafenamide (E/C/F/TAF) 150/150/200/10 mg fixed dose combination (FDC) tablets administered orally once daily with food for 48 weeks
- ABC/3TC+3rd Agent: Abacavir/lamivudine (ABC/3TC) 600/300 mg tablets plus a third antiretroviral agent administered orally once daily for 24 weeks followed by a delayed switch to E/C/F/TAF FDC
Period: Overall Study
Arm/Group | E/C/F/TAF | ABC/3TC+3rd Agent
Started | 183 | 92
Completed | 171 | 88
Not Completed | 12 | 4
Not completed — Adverse Event | 5 | 1
Not completed — Investigator's Discretion | 1 | 0
Not completed — Non-Compliance with Study Drug | 1 | 0
Not completed — Withdrew Consent | 2 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Randomized but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who took at least 1 dose of E/C/F/TAF or ABC/3TC+3rd Agent (on or after Day 1).
Groups:
- E/C/F/TAF: E/C/F/TAF (150/150/200/10 mg) FDC tablets administered orally once daily with food for 48 weeks
- ABC/3TC+3rd Agent: ABC/3TC (600/300 mg) tablets plus a third antiretroviral agent administered orally once daily for 24 weeks followed by a delayed switch to E/C/F/TAF FDC
- Total: Total of all reporting groups
Arm/Group | E/C/F/TAF | ABC/3TC+3rd Agent | Total
Number analyzed (Participants) | 183 | 91 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (11.6) | 49 (10.7) | 49 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 17 | 44
  Male | 156 | 74 | 230
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 1 | 6
  Black | 27 | 15 | 42
  White | 150 | 75 | 225
  Other | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 16 | 43
  Not Hispanic or Latino | 155 | 73 | 228
  Not Permitted | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 19 | 55
  Italy | 43 | 16 | 59
  United Kingdom | 2 | 1 | 3
  France | 40 | 23 | 63
  Germany | 6 | 2 | 8
  Spain | 56 | 30 | 86
HIV-1 RNA Categories [Count of Participants; unit: Participants]
  < 50 copies/mL | 177 | 91 | 268
  50 ≥ copies/mL | 6 | 0 | 6
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 701 (280.1) | 753 (312.8) | 718 (291.8)
CD4 Cell Count Category [Count of Participants; unit: Participants]
  ≥ 50 to < 200 cells/µL | 2 | 0 | 2
  ≥ 200 to < 350 cells/µL | 11 | 7 | 18
  ≥ 350 to < 500 cells/µL | 30 | 13 | 43
  ≥ 500 cells/µL | 140 | 71 | 211

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have HIV-1 RNA < 50 Copies/mL as Defined by the FDA Snapshot Algorithm at Week 24
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Full Analysis Set: participants who were randomized and received at least one dose of study drug (either E/C/F/TAF or ABC/3TC+3rd agent on or after Day 1).
Measure: Number; unit: percentage of participants
Groups:
- Delayed E/C/F/TAF: Participants in 'ABC/3TC+3rd agent' group who switched to E/C/F/TAF group at Week 24 received E/C/F/TAF (150/150/200/10 mg) FDC tablets orally once daily with food.
Arm/Group | E/C/F/TAF | ABC/3TC+3rd Agent | Delayed E/C/F/TAF
Number analyzed (Participants) | 183 | 91 | 89
percentage of participants | 93.4 | 97.8 | 96.6
Statistical Analysis 1: Comparison: E/C/F/TAF vs ABC/3TC+3rd Agent; Test type: Non-Inferiority — With 200 participants randomized to switch to the E/C/F/TAF FDC group at Day 1 and 100 participants randomized to the ABC/3TC+3rd Agent group at Week 24, the lower limit of the observed one sided 97.5% confidence interval was expected to be greater than -0.120 (ie, non-inferiority margin of 12%) with > 90% power when the percentage of responders in both treatment groups for the primary endpoint is at least 90% at Week 24; p = 0.15, Fisher Exact; Difference in Percentages = -4.4, 95% CI 2-sided [-9.4 to 1.9]

2. Secondary Outcome: Percentage of Participants Who Have HIV-1 RNA < 50 Copies/mL as Defined by the FDA Snapshot Algorithm at Week 12
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at week 12 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | ABC/3TC+3rd Agent | Delayed E/C/F/TAF
Number analyzed (Participants) | 183 | 91 | 89
percentage of participants | 95.1 | 98.9 | 96.6
Statistical Analysis 1: Comparison: E/C/F/TAF vs ABC/3TC+3rd Agent; Test type: Non-Inferiority — With 200 participants randomized to switch to the E/C/F/TAF FDC group at Day 1 and 100 participants randomized to the delayed switch group at Week 12, the lower limit of the observed one sided 97.5% confidence interval will be expected to be greater than -0.120 (ie, non-inferiority margin of 12%) with > 90% power when the percentage of responders in both treatment groups for the primary endpoint is at least 90% at Week 12; p = 0.17, Fisher Exact; Difference in Percentages = -3.8, 95% CI 2-sided [-8.3 to 1.6]

3. Secondary Outcome: Percentage of Participants Who Have HIV-1 RNA < 50 Copies/mL as Defined by the FDA Snapshot Algorithm at Week 48
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Only the participants who were randomized to E/C/F/TAF group were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF
Number analyzed (Participants) | 183
percentage of participants | 86.9

4. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | E/C/F/TAF | ABC/3TC+3rd Agent | Delayed E/C/F/TAF
Number analyzed (Participants) | 169 | 90 | 86
cells/µL | -28 (161.4) | 8 (192.9) | -23 (201.7)
Statistical Analysis 1: Comparison: E/C/F/TAF vs ABC/3TC+3rd Agent; Test type: Other; p = 0.11, ANOVA; Difference in least square mean = -36, 95% CI 2-sided [-80 to 9]

5. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the E/C/F/TAF group with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | E/C/F/TAF
Number analyzed (Participants) | 156
cells/µL | -32 (147.1)

ADVERSE EVENTS:
Time Frame: Up to 48 weeks plus 30 days
Description: The reported percentages in the Adverse Events table were not adjusted for the different durations in adverse events (AE) collection. By study design, the AE collection time frame for the treatment groups was as follows:
  * E/C/F/TAF group = 48 weeks plus 30 days
  * ABC/3TC+3rd Agent = 24 weeks
  * Delayed E/C/F/TAF group = 24 weeks plus 30 days
Groups:
- All E/C/F/TAF: Adverse events in this reporting group include those that occurred any time during the study by participants while receiving E/C/F/TAF.
  Participants received E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily with food.
Arm/Group | E/C/F/TAF | ABC/3TC+3rd Agent | Delayed E/C/F/TAF | All E/C/F/TAF
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/91 | 0/89 | 0/272
Serious Adverse Events (participants affected / at risk) | 12/183 | 1/91 | 4/89 | 16/272
Other Adverse Events (participants affected / at risk) | 71/183 | 21/91 | 17/89 | 88/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TAF (N=183) | ABC/3TC+3rd Agent (N=91) | Delayed E/C/F/TAF (N=89) | All E/C/F/TAF (N=272)
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 1
Hepatitis A (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 2
Device dislocation (Product Issues) | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TAF (N=183) | ABC/3TC+3rd Agent (N=91) | Delayed E/C/F/TAF (N=89) | All E/C/F/TAF (N=272)
Diarrhoea (Gastrointestinal disorders) | 19 | 3 | 4 | 23
Asthenia (General disorders) | 10 | 1 | 0 | 10
Upper respiratory tract infection (Infections and infestations) | 12 | 5 | 1 | 13
Vitamin D deficiency (Metabolism and nutrition disorders) | 13 | 6 | 0 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 2 | 8 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 6 | 2 | 8
Headache (Nervous system disorders) | 15 | 4 | 4 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol: Original (2015-07-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT02605954/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT02605954/Prot_001.pdf
  • Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT02605954/SAP_002.pdf